CLINICAL TRIAL: NCT03657849
Title: Evaluation of 19-gauge vs 21-gauge EBUS TBNA in Assessing Thoracic Lymphadenopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A18-177
Record Dates: First submitted 2018-07-31; First posted 2018-09-05 (Actual); Results first posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2019-08

CONDITIONS: Enlarged Lymph Nodes (Excluding Infective)
MeSH Terms: conditions — Lymphadenopathy

STUDY DESIGN:
Intervention Model Description: Prospective diagnostic accuracy study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Sampling with 19-gauge and 21-gauge (Experimental): All patients will be allocated to the same arm. All patients will have EBUS TBNA done with both 19-gauge and 21-gauge needles during the procedure.
  Interventions: Device: EBUS TBNA

INTERVENTIONS:
Device: EBUS TBNA — All patients undergo EBUS TBNA with two needle sizes

SUMMARY:
This study compares the yield of 19-gauge needles vs 21-gauge needles during EBUS TBNA procedures.

DETAILED DESCRIPTION:
Endobronchial ultrasound-guided transbronchial needle aspirate (EBUS-TBNA) is a technique used to take samples of body tissue inside the chest without having to undergo an operation.

During this procedure, a special telescope (called a bronchoscope) is inserted through the mouth into the airways. Ultrasound technology allows the doctor to see the structures just outside the airway. By being able to see the structures outside the airway, the doctor is able to safely pass a fine needle through the airway to take samples of abnormal tissue.

EBUS-TBNA is used to take samples of tissue from the mediastinum. The mediastinum is the part of the chest between the lungs, and contains the heart, gullet, windpipe and lymph nodes. This area of the body is usually difficult to access without open surgery, hence the use of EBUS-TBNA. EBUS-TBNA may be used to investigate enlarged lymph nodes. This may be due to tuberculosis, sarcoidosis or cancer.

Currently, smaller 21-gauge and larger 19-gauge needles are used during the EBUS-TBNA procedure at Regions Hospital. The purpose of this study is to find out which needle is better in finding the explanation for the enlarged lymph nodes, and any follow up procedures that may be necessary if the investigators are unable to get enough tissue during the EBUS-TBNA procedure (surgical sampling, radiological sampling, and/or follow-up imaging).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able to provide informed consent
* Referred for EBUS TBNA sampling at Regions Hospital

Exclusion Criteria:

* On therapeutic warfarin, Plavix, or ticagrelor in the past 5 days
* INR>1.8 or platelets <50K

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Firas S Elmufdi, MBBS, Principal Investigator — Regions Hospital
Locations (1):
- Regions Hospital, Saint Paul, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 consecutive patients referred for EBUS-TBNA sampling between July 2018 and January 2019 were enrolled after providing written consent.
Pre-assignment Details: A total of 144 lymph nodes were sampled from the 60 enrolled. Of these, 3 lymph nodes were excluded from analysis due to protocol deviations (two were only sampled with one needle and the third underwent one pass before the provider decided to change sites).
Units Other Than Participants: Lymph nodes
Period: Overall Study
Arm/Group | Sampling With 19-gauge and 21-gauge
Started | 60; 144 Lymph nodes
Completed | 60; 141 Lymph nodes (Although 3 lymph nodes were excluded from analysis, at least 1 lymph node from each participant was included. The 3 excluded lymph nodes were removed due to protocol deviations related to sampling.)
Not Completed | 0; 3 Lymph nodes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Lymph nodes
Arm/Group | Sampling With 19-gauge and 21-gauge
Number analyzed (Participants) | 60
Number analyzed (Lymph nodes) | 141
Age, Customized [Count of Participants; unit: Participants]
  Age Distribution: Patients < 18 | 0
  Age Distribution: Patients >/= 18 | 60
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 30
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Yield
Description: Diagnostic yield refers to the proportion of tissue samples collected by each needle (19 gauge vs 21 gauge) that were of sufficient quantity and quality to yield (i.e. produce) an accurate diagnosis for the patient's enlarged lymph nodes. Characterization of diagnostic category (true positive, true negative, false negative, false positive) were made by comparing the patient's presumed diagnosis/initial indication for presentation in comparison to their final diagnosis as determined by a combination of pathological findings of EBUS-TBNA, follow up imaging, surgical sampling, or clinical follow up. The diagnostic yield of each needles was reported as a ratio of true positives and true negatives added together, divided by the total number of lymph nodes sampled (141).
  Diagnostic yield of 19-gauge needle: 89.4% Diagnostic yield of 21-gauge needled: 88.7%
Time Frame: 6 months
Population: All 141 lymph nodes included in the final analysis were sampled by both the 19-guage and 21-guage needle. Participants were randomized to a particular ordering of the needles (either the 19-gauge or 21-guage needle would be used to sample lymph nodes sites first, followed by which ever remaining needle had not been used).
Measure: Count of Units; unit: lymph nodes
Units Other Than Participants: lymph nodes
Groups:
- 19-Gauge Needle; 21-Gauge Needle: All lymph nodes included in the final analysis were sampled with the 19-gauge and 21-gauge needles. Results will be reported per intervention.
Arm/Group | 19-Gauge Needle | 21-Gauge Needle
Number analyzed (Participants) | 60 | 60
Number analyzed (lymph nodes) | 141 | 141
lymph nodes
  True Positives | 69 | 68
  True Negatives | 57 | 57
  False Negatives + False Positives (Not included in calculation of diagnostic yield) | 15 | 16

2. Primary Outcome: Diagnostic Yield
Description: Diagnostic yield refers to the proportion of tissue samples collected by each needle (19 gauge vs 21 gauge) that were of sufficient quantity and quality to yield (i.e. produce) an accurate diagnosis for the patient's enlarged lymph nodes. Characterization of diagnostic category (true positive, true negative, false negative, false positive) were made by comparing the patient's presumed diagnosis/initial indication for presentation in comparison to their final diagnosis as determined by a combination of pathological findings of EBUS-TBNA, follow up imaging, surgical sampling, or clinical follow up. The diagnostic yield of each needles was reported as a ratio of true positives and true negatives added together, divided by the total number of lymph nodes sampled (141).
Time Frame: 6 months
Measure: Count of Units; unit: lymph nodes
Units Other Than Participants: lymph nodes
Arm/Group | 19-Gauge Needle | 21-Gauge Needle
Number analyzed (Participants) | 60 | 60
Number analyzed (lymph nodes) | 141 | 141
lymph nodes | 126 | 125

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from the time the patient signed the consent form (i.e. immediately prior to the Endobronchial ultrasound (EBUS) transbronchial needle aspiration (TBNA) procedure), to the point at which the results of the confirmed and a final diagnosis was reported to the participant. Although the follow-up period varied by participant, the average length of time over which adverse events tracked and reported was 6 months.
Description: Adverse events could not be reported per intervention (i.e., 19G versus 21G). The "passes" made on each lymph node using both gauge needles occurred in such close proximity to one other (on the order of seconds) that it would be impossible to determine what adverse events were related to which gauge needle. The adverse events listed relate to the overall bronchoscopic-biopsy procedure rather than to the size of the needle used during the biopsies.
Groups:
- 19-Gauge Needle Used First: Patients in this arm had their lymph nodes sampled with the 19-gauge needle first, followed by the 21-gauge needle.
  All patients were sampled by both needles; randomization and group arm assignment controlled for the order in which the needles were used.
- 21-Gauge Needle Used First: Patients in this arm had their lymph nodes sampled with the 21-gauge needle first, followed by the 19-gauge needle.
  All patients were sampled by both needles; randomization and group arm assignment controlled for the order in which the needles were used.
Arm/Group | 19-Gauge Needle Used First | 21-Gauge Needle Used First
All-Cause Mortality (participants affected / at risk) | 0/30 | 1/30
Serious Adverse Events (participants affected / at risk) | 1/30 | 2/30
Other Adverse Events (participants affected / at risk) | 3/30 | 4/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 19-Gauge Needle Used First (N=30) | 21-Gauge Needle Used First (N=30)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Patient died during follow-up period as a result of respiratory failure secondary to underlying small cell lung cancer (a condition present at baseline).
acute hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Patient experienced a bronchospasm as a result of bronchoscopy, resulting in acute hypoxic respiratory failure that was treated with nebulizers and BiPAP.
Missing 19-guage needle spring (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — During EBUS procedure it was noted that there was the lost of 19 gauge needle spring. This was categorized as not severe, as the spring has not been noted in the patient x-rays or during evaluation of the patient.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 19-Gauge Needle Used First (N=30) | 21-Gauge Needle Used First (N=30)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — Three patients noted to have mild hypoxia following procedure. Two resolved; one patient left against medical advise after being asked to stay under observation for low O2 sats
Blood clot (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 — small airway clots noted following bronchoscopy procedure, noted to be mild.
Hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) — Patient experienced hypotension as a result of sedation used for procedure; resolved with nalaxone.
Nausea/Vertigo (Gastrointestinal disorders) | 0 (0) | 1 (1) — patient has history of nausea and vertigo; experienced symptoms after the procedure under investigation was completed.
Bleeding (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — patient Experienced minor bleeding at the site and time of procedure.
poor ventilation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Patient experienced violent coughing during first attempt at bronchoscopy. Additional sedation was given to prevent coughing, but the patient experienced poor ventilation and a "jaw thrust" was implemented for10 seconds during the procedure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT03657849/Prot_SAP_000.pdf